CLINICAL TRIAL: NCT01924806
Title: A Pilot Study of the WoundWand™ Debridement Device on Infection Prevention
Acronym: WoundWand
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lower than expected accrual rate and desire to reassess overall study strategy.
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WW-2013-02
Record Dates: First submitted 2013-08-13; First posted 2013-08-19 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Lower Leg Wound
Keywords: debridement; post-debridement; infection; prevention; wound; wound tissue; wound management; WoundWand; wound size reduction; wound bed debridement; WoundWand Debridement Device; chronic wound; delayed healing; cellular senescence; acute wound; diabetic foot ulcer; venous leg ulcers; radiofrequency debridement; necrotic tissue; wound healing; skin
MeSH Terms: conditions — Infections; Wounds and Injuries; Diabetic Foot

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- WoundWand™ Debridement Device (Active Comparator): Group I - Coblator IQTM Controller plus WoundWandTM Debridement Device. Electrical energy that removes necrotic, ischemic, and/or infected tissue within a wound.
  Interventions: Device: WoundWand™ Debridement Device
- Standard of Care sharp debridement (Active Comparator): Group II - Standard of Care (SoC) surgical (sharp) debridement. Sharp instruments that remove necrotic, ischemic, and/or infected tissue within a wound.
  Interventions: Device: Standard of Care sharp debridement

INTERVENTIONS:
Device: WoundWand™ Debridement Device — Group I - Electrical energy that removes necrotic, ischemic, and/or infected tissue within a wound
  Arms: WoundWand™ Debridement Device
Device: Standard of Care sharp debridement — Group II - Sharp instruments that remove necrotic, ischemic, and/or infected tissue within a wound
  Arms: Standard of Care sharp debridement

SUMMARY:
A Pilot Study of the WoundWand™ Debridement Device on Infection Prevention

DETAILED DESCRIPTION:
The primary aim of this pilot study is to investigate differences in bacterial content of the study wound that may impact upon infection rates following debridement with the WoundWand Debridement Device or Standard of Care (SoC) surgical (sharp) debridement. Additionally, the clinical investigation will evaluate reduction in wound size post-debridement and gather Health Economic data relating to wound bed debridement with the WoundWand Debridement Device or SoC.

ELIGIBILITY:
Inclusion Criteria

Subjects who meet the following criteria may be included in the clinical investigation, if they present with ALL of the following:

1. Subject is able to understand the evaluation and willing to consent and comply with all post-debridement visits and procedures
2. Age 18 years and older. Subjects may be of either sex and of any race or skin type
3. Subjects fulfilling any one or all of the following criteria:

   1. chronic wound(s) below the level of the knee, defined by delayed healing or cellular senescence
   2. acute wound(s) as a result of a surgical procedure, laceration, abrasion or trauma
   3. diabetic foot ulcer(s)
   4. subjects with venous leg ulcers below the knee on the leg or foot with one or more documented failure of maximal medical therapy for their study wound >30 days such as compression bandages (low elasticity, elastic, multilayered, elastic and non elastic compression)
4. Subjects with the following lab results within 30 days of treatment:

   1. serum albumin level >20g/L
   2. clinically non significant results of liver function test (LFTs), serum glucose and complete blood count (CBC) with differential
5. Subjects with a Braden Score ≥13-14 (Moderate Risk)
6. Subjects with adequate arterial blood flow [Ankle-Brachial Index (ABI) >0.75]

Exclusion Criteria

Subjects will be excluded from the clinical investigation, if they present with ANY of the following:

1. Subjects that have tunneling wounds
2. Subject presents with an active infection in the study wound, as defined by purulence and:

   1. Fever and leukocytosis

      OR any TWO of the following:
   2. Malodor, pain or tenderness, warmth, erythema, induration, swelling, lymphangitis
3. Infected bone diagnosed by imaging modality (e.g., Magnetic Resonance Imaging (MRI) and/or radiographic images)
4. Subjects whose study wound does not require debridement
5. Cardiac pacemaker or other electronic implant(s)
6. Subjects with irradiate, burn or ischaemic wounds or history of keloids
7. Subjects with vasculitis, non-reconstructive peripheral vascular disease, pyoderma gangrenosum, renal failure or lymphoedema
8. Subjects with uncontrolled bleeding disorder (PT/PTT) and coagulopathy (including those with hemophilia)
9. Subjects taking treatment with any of the following:

   1. Systemic corticosteroids
   2. Immunosuppressive agent(s)
   3. Chemotherapy or Radiation therapy
10. Subjects deemed to require biologic dressing/ skin substitute
11. Terminally ill subjects
12. Subjects that have an immunodeficiency disorder that interferes with wound healing, including Acquired Immunodeficiency Syndrome (AIDS) or know to be infected with Human Immunodeficiency Virus (HIV)
13. Subjects that have chronic skin conditions such as psoriasis, etc.
14. Subjects that reside in a nursing home
15. Subject is physically or mentally compromised (e.g., currently being treated for a psychiatric disorder, senile dementia, Alzheimer's disease, etc.) to the extent that the Investigator judges the subject to be unable or unlikely to remain compliant
16. Subject is pregnant and/or intending to become pregnant during this clinical investigation period
17. Subject has documented evidence of a history (e.g. liver testing) of drug/alcohol abuse within the 12 months prior to enrollment for clinical investigation entry
18. Subject is excluded if they have received an investigational therapy or approved therapy for investigational use within 30 days of surgery
19. Subject is excluded if planning to participate in another research study during the follow-up phase of this study or 84 days after study completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-03-04 (Actual); Primary Completion 2015-02-09 (Actual); Study Completion 2015-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luc Teot, M.D. Phd., Principal Investigator — Hopital Lapeyronie; Beate Hanson, MD, PhD, Study Chair — Vice President, Global Clinical Strategy
Locations (2):
- Hopital Lapeyronie, Montpellier, France
- Manchester Diabetes Centre, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty (60) subjects were to be randomized in a 1:1 ratio. A total of 11 subjects were enrolled at 1 investigative site by 2 investigators.
Pre-assignment Details: Overall, 9 subjects received treatment for a total of 9 wounds treated. Two of the enrolled subjects, discontinued prior to treatment.
Units Other Than Participants: Wounds
Groups:
- WoundWand™ Debridement Device: WoundWand™ Debridement Device: Group I - Electrical energy that removes necrotic, ischemic, and/or infected tissue within a wound. ArthroCare developed COBLATION® technology, which uses a controlled, non-heat drive process (i.e., radiofrequency energy) to gently and precisely dissolve soft tissue, thereby minimizing damage to healthy tissue. ArthroCare adapted this technology for use in wound debridement via the WoundWand Debridement Device.
- Standard of Care Sharp Debridement: Standard of Care sharp debridement: Group II - Sharp instruments that remove necrotic, ischemic, and/or infected tissue within a wound. Surgical or sharp debridement is one of the methods commonly used to remove necrotic tissue from non-healing and difficult-to-heal chronic wounds. Surgical debridement requires sterile instruments and a qualified clinician in addition to general or local anesthesia.
Period: Overall Study
Arm/Group | WoundWand™ Debridement Device | Standard of Care Sharp Debridement
Started | 5; 5 Wounds | 4; 4 Wounds
Completed | 3; 3 Wounds | 3; 3 Wounds
Not Completed | 2; 2 Wounds | 1; 1 Wounds
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Population: All randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | WoundWand™ Debridement Device | Standard of Care Sharp Debridement | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (8.6) | 68.8 (13.6) | 67.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 5 | 4 | 9
Etiology of Study Wound [Count of Participants; unit: Participants]
  Pressure | 2 | 2 | 4
  Pressure and Neuropathy | 0 | 1 | 1
  Infection | 1 | 0 | 1
  Infection, Trauma and Neuropathy | 0 | 1 | 1
  Laceration | 0 | 0 | 0
  Abrasion | 0 | 0 | 0
  Trauma | 0 | 0 | 0
  Surgical Procedure | 0 | 0 | 0
  Surgical Procedure and Underlying Condition | 1 | 0 | 1
  Vascular Insufficiency | 1 | 0 | 1
  Neuropathy | 0 | 0 | 0
  Underlying Condition | 0 | 0 | 0
  Other | 0 | 0 | 0
Type of Wound [Count of Participants; unit: Participants]
  Chronic | 0 | 1 | 1
  Chronic and Diabetic Foot Ulcer | 0 | 2 | 2
  Acute | 0 | 0 | 0
  Diabetic Foot Ulcer | 5 | 1 | 6
  Venous Leg Ulcer | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Bacterial Diversity and Number of Bacteria Present in the Wound
Description: Primary endpoint was to determine bacterial diversity and number of bacteria present in the study wound at 4 weeks post- debridement using either WoundWand Debridement Device or Standard of Care. Punch biopsies were performed per standard practice to quantify the type and amount of bacteria present in wounds debrided with either Standard of Care Sharp Debridement or WoundWand Debridement Device. Debridement of contaminated tissue is essential to prevent wound infection, promote healing, and provide a neat wound edge for the prevention of scaring.
  A 3-4 mm punch biopsy for quantitative tissue culture (i.e. bacterial content) will be collected from the study wound site immediately pre- and post-debridement and at Week 4. The punch biopsy will be performed per standard practice and if required, utilizing the appropriate analgesia [e.g. general, local (e.g. 1% lidocaine with epinephrine)]. Quantitative tissue culture will be completed according to the laboratory's standard procedures
Time Frame: Day 1 (immediately pre- and post-debridement) and 4 weeks post-debridement
Population: All treated subjects
Measure: Number; unit: Log^10 CFU/g
Arm/Group | WoundWand™ Debridement Device | Standard of Care Sharp Debridement
Number analyzed (Participants) | 5 | 4
Log^10 CFU/g
  Subject 02-001 - Total Aerobes/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-001 - Total Aerobes/Pre | 7.74 |
  02-001 - Total Aerobes/Post: number analyzed (Participants) | 1 | 0
  02-001 - Total Aerobes/Post | 7.25 |
  02-001 - Total Aerobes/Week 4: number analyzed (Participants) | 1 | 0
  02-001 - Total Aerobes/Week 4 | 6.29 |
  Subject 02-002 - Total Aerobes/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-002 - Total Aerobes/Pre |  | 8.37
  02-002 - Total Aerobes/Post: number analyzed (Participants) | 0 | 1
  02-002 - Total Aerobes/Post |  | 7.05
  02-002 - Total Aerobes/Week 4: number analyzed (Participants) | 0 | 1
  02-002 - Total Aerobes/Week 4 |  | 5.31
  Subject 02-003 - Total Aerobes/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-003 - Total Aerobes/Pre | 9.14 |
  02-003 - Total Aerobes/Post: number analyzed (Participants) | 1 | 0
  02-003 - Total Aerobes/Post | 4.38 |
  02-003 - Total Aerobes/Week 4: number analyzed (Participants) | 1 | 0
  02-003 - Total Aerobes/Week 4 | 6.67 |
  Subject 02-004 - Total Aerobes/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-004 - Total Aerobes/Pre |  | 5.99
  02-004 - Total Aerobes/Post: number analyzed (Participants) | 0 | 1
  02-004 - Total Aerobes/Post |  | 4.91
  02-004 - Total Aerobes/Week 4: number analyzed (Participants) | 0 | 1
  02-004 - Total Aerobes/Week 4 |  | 7.70
  Subject 02-005 - Total Aerobes/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-005 - Total Aerobes/Pre |  | 8.46
  02-005 - Total Aerobes/Post: number analyzed (Participants) | 0 | 1
  02-005 - Total Aerobes/Post |  | 6.75
  02-005 - Total Aerobes/Week 4: number analyzed (Participants) | 0 | 1
  02-005 - Total Aerobes/Week 4 |  | 6.38
  Subject 02-007 - Total Aerobes/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-007 - Total Aerobes/Pre | 7.42 |
  02-007 - Total Aerobes/Post: number analyzed (Participants) | 1 | 0
  02-007 - Total Aerobes/Post | 5.12 |
  02-007 - Total Aerobes/Week 4: number analyzed (Participants) | 1 | 0
  02-007 - Total Aerobes/Week 4 | 8.08 |
  Subject 02-008 - Total Aerobes/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-008 - Total Aerobes/Pre |  | 7.84
  02-008 - Total Aerobes/Post: number analyzed (Participants) | 0 | 1
  02-008 - Total Aerobes/Post |  | 7.41
  02-008 - Total Aerobes/Week 4: number analyzed (Participants) | 0 | 1
  02-008 - Total Aerobes/Week 4 |  | 4.09
  Subject 02-009 - Total Aerobes/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-009 - Total Aerobes/Pre | 6.90 |
  02-009 - Total Aerobes/Post: number analyzed (Participants) | 1 | 0
  02-009 - Total Aerobes/Post | 4.41 |
  02-009 - Total Aerobes/Week 4: number analyzed (Participants) | 1 | 0
  02-009 - Total Aerobes/Week 4 | 8.56 |
  Subject 02-010 - Total Aerobes/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-010 - Total Aerobes/Pre | 7.30 |
  02-010 - Total Aerobes/Post: number analyzed (Participants) | 1 | 0
  02-010 - Total Aerobes/Post | 7.24 |
  02-010 - Total Aerobes/Week 4: number analyzed (Participants) | 1 | 0
  02-010 - Total Aerobes/Week 4 | 8.79 |
  Subject 02-001 - Total Gram Positive Anaerobes/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-001 - Total Gram Positive Anaerobes/Pre | 7.66 |
  02-001 - Total Gram + Anaerobes/Post: number analyzed (Participants) | 1 | 0
  02-001 - Total Gram + Anaerobes/Post | 5.25 |
  02-001 - Total Gram + Anaerobes/Week 4: number analyzed (Participants) | 1 | 0
  02-001 - Total Gram + Anaerobes/Week 4 | 5.66 |
  Subject 02-002 - Total Gram Positive Anaerobes/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-002 - Total Gram Positive Anaerobes/Pre |  | 8.50
  02-002 - Total Gram + Anaerobes/Post: number analyzed (Participants) | 0 | 1
  02-002 - Total Gram + Anaerobes/Post |  | 7.05
  02-002 - Total Gram + Anaerobes/Week 4: number analyzed (Participants) | 0 | 1
  02-002 - Total Gram + Anaerobes/Week 4 |  | 3.83
  Subject 02-003 - Total Gram Positive Anaerobes/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-003 - Total Gram Positive Anaerobes/Pre | 8.66 |
  02-003 - Total Gram + Anaerobes/Post: number analyzed (Participants) | 1 | 0
  02-003 - Total Gram + Anaerobes/Post | 3.36 |
  02-003 - Total Gram + Anaerobes/Week 4: number analyzed (Participants) | 1 | 0
  02-003 - Total Gram + Anaerobes/Week 4 | 7.60 |
  Subject 02-004 - Total Gram Positive Anaerobes/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-004 - Total Gram Positive Anaerobes/Pre |  | 5.02
  02-004 - Total Gram + Anaerobes/Post: number analyzed (Participants) | 0 | 1
  02-004 - Total Gram + Anaerobes/Post |  | 3.80
  02-004 - Total Gram + Anaerobes/Week 4: number analyzed (Participants) | 0 | 1
  02-004 - Total Gram + Anaerobes/Week 4 |  | 6.43
  Subject 02-005 - Total Gram Positive Anaerobes/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-005 - Total Gram Positive Anaerobes/Pre |  | 7.42
  02-005 - Total Gram + Anaerobes/Post: number analyzed (Participants) | 0 | 1
  02-005 - Total Gram + Anaerobes/Post |  | 5.58
  02-005 - Total Gram + Anaerobes/Week 4: number analyzed (Participants) | 0 | 1
  02-005 - Total Gram + Anaerobes/Week 4 |  | 4.56
  Subject 02-007 - Total Gram Positive Anaerobes/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-007 - Total Gram Positive Anaerobes/Pre | 5.28 |
  02-007 - Total Gram + Anaerobes/Post: number analyzed (Participants) | 1 | 0
  02-007 - Total Gram + Anaerobes/Post | 3.29 |
  02-007 - Total Gram + Anaerobes/Week 4: number analyzed (Participants) | 1 | 0
  02-007 - Total Gram + Anaerobes/Week 4 | 3.92 |
  Subject 02-008 - Total Gram Positive Anaerobes/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-008 - Total Gram Positive Anaerobes/Pre |  | 7.61
  02-008 - Total Gram + Anaerobes/Post: number analyzed (Participants) | 0 | 1
  02-008 - Total Gram + Anaerobes/Post |  | 7.41
  02-008 - Total Gram + Anaerobes/Week 4: number analyzed (Participants) | 0 | 1
  02-008 - Total Gram + Anaerobes/Week 4 |  | 0.00
  Subject 02-009 - Total Gram Positive Anaerobes/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-009 - Total Gram Positive Anaerobes/Pre | 4.28 |
  02-009 - Total Gram + Anaerobes/Post: number analyzed (Participants) | 1 | 0
  02-009 - Total Gram + Anaerobes/Post | 0.00 |
  02-009 - Total Gram + Anaerobes/Week 4: number analyzed (Participants) | 1 | 0
  02-009 - Total Gram + Anaerobes/Week 4 | 8.70 |
  Subject 02-010 - Total Gram Positive Anaerobes/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-010 - Total Gram Positive Anaerobes/Pre | 4.30 |
  02-010 - Total Gram + Anaerobes/Post: number analyzed (Participants) | 1 | 0
  02-010 - Total Gram + Anaerobes/Post | 3.15 |
  02-010 - Total Gram + Anaerobes/Week 4: number analyzed (Participants) | 1 | 0
  02-010 - Total Gram + Anaerobes/Week 4 | 7.66 |
  Subject 02-001 - Total Gram Negative Anaerobes/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-001 - Total Gram Negative Anaerobes/Pre | 6.98 |
  02-001 - Total Gram - Anaerobes/Post: number analyzed (Participants) | 1 | 0
  02-001 - Total Gram - Anaerobes/Post | 3.21 |
  02-001 - Total Gram - Anaerobes/Week 4: number analyzed (Participants) | 1 | 0
  02-001 - Total Gram - Anaerobes/Week 4 | 4.80 |
  Subject 02-002 - Total Gram Negative Anaerobes/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-002 - Total Gram Negative Anaerobes/Pre |  | 7.30
  02-002 - Total Gram - Anaerobes/Post: number analyzed (Participants) | 0 | 1
  02-002 - Total Gram - Anaerobes/Post |  | 5.57
  02-002 - Total Gram - Anaerobes/Week 4: number analyzed (Participants) | 0 | 1
  02-002 - Total Gram - Anaerobes/Week 4 |  | 4.75
  Subject 02-003 - Total Gram Negative Anaerobes/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-003 - Total Gram Negative Anaerobes/Pre | 8.90 |
  02-003 - Total Gram - Anaerobes/Post: number analyzed (Participants) | 1 | 0
  02-003 - Total Gram - Anaerobes/Post | 3.70 |
  02-003 - Total Gram - Anaerobes/Week 4: number analyzed (Participants) | 1 | 0
  02-003 - Total Gram - Anaerobes/Week 4 | 0.00 |
  Subject 02-004 - Total Gram Negative Anaerobes/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-004 - Total Gram Negative Anaerobes/Pre |  | 0.00
  02-004 - Total Gram - Anaerobes/Post: number analyzed (Participants) | 0 | 1
  02-004 - Total Gram - Anaerobes/Post |  | 0.00
  02-004 - Total Gram - Anaerobes/Week 4: number analyzed (Participants) | 0 | 1
  02-004 - Total Gram - Anaerobes/Week 4 |  | 5.88
  Subject 02-005 - Total Gram Negative Anaerobes/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-005 - Total Gram Negative Anaerobes/Pre |  | 6.54
  02-005 - Total Gram - Anaerobes/Post: number analyzed (Participants) | 0 | 1
  02-005 - Total Gram - Anaerobes/Post |  | 5.59
  02-005 - Total Gram - Anaerobes/Week 4: number analyzed (Participants) | 0 | 1
  02-005 - Total Gram - Anaerobes/Week 4 |  | 6.30
  Subject 02-007 - Total Gram Negative Anaerobes/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-007 - Total Gram Negative Anaerobes/Pre | 7.54 |
  02-007 - Total Gram - Anaerobes/Post: number analyzed (Participants) | 1 | 0
  02-007 - Total Gram - Anaerobes/Post | 5.13 |
  02-007 - Total Gram - Anaerobes/Week 4: number analyzed (Participants) | 1 | 0
  02-007 - Total Gram - Anaerobes/Week 4 | 7.89 |
  Subject 02-008 - Total Gram Negative Anaerobes/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-008 - Total Gram Negative Anaerobes/Pre |  | 3.31
  02-008 - Total Gram - Anaerobes/Post: number analyzed (Participants) | 0 | 1
  02-008 - Total Gram - Anaerobes/Post |  | 0.00
  02-008 - Total Gram - Anaerobes/Week 4: number analyzed (Participants) | 0 | 1
  02-008 - Total Gram - Anaerobes/Week 4 |  | 0.00
  Subject 02-009 - Total Gram Negative Anaerobes/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-009 - Total Gram Negative Anaerobes/Pre | 5.82 |
  02-009 - Total Gram - Anaerobes/Post: number analyzed (Participants) | 1 | 0
  02-009 - Total Gram - Anaerobes/Post | 3.96 |
  02-009 - Total Gram - Anaerobes/Week 4: number analyzed (Participants) | 1 | 0
  02-009 - Total Gram - Anaerobes/Week 4 | 3.59 |
  Subject 02-010 - Total Gram Negative Anaerobes/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-010 - Total Gram Negative Anaerobes/Pre | 5.73 |
  02-010 - Total Gram - Anaerobes/Post: number analyzed (Participants) | 1 | 0
  02-010 - Total Gram - Anaerobes/Post | 6.07 |
  02-010 - Total Gram - Anaerobes/Week 4: number analyzed (Participants) | 1 | 0
  02-010 - Total Gram - Anaerobes/Week 4 | 8.62 |
  Subject 02-001 - Total Staphylococci/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-001 - Total Staphylococci/Pre | 7.11 |
  02-001 - Total Staph/Post: number analyzed (Participants) | 1 | 0
  02-001 - Total Staph/Post | 4.56 |
  02-001 - Total Staph/Week 4: number analyzed (Participants) | 1 | 0
  02-001 - Total Staph/Week 4 | 0.00 |
  Subject 02-002 - Total Staphylococci/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-002 - Total Staphylococci/Pre |  | 6.39
  02-002 - Total Staph/Post: number analyzed (Participants) | 0 | 1
  02-002 - Total Staph/Post |  | 5.92
  02-002 - Total Staph/Week 4: number analyzed (Participants) | 0 | 1
  02-002 - Total Staph/Week 4 |  | 0.00
  Subject 02-003 - Total Staphylococci/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-003 - Total Staphylococci/Pre | 8.75 |
  02-003 - Total Staph/Post: number analyzed (Participants) | 1 | 0
  02-003 - Total Staph/Post | 4.38 |
  02-003 - Total Staph/Week 4: number analyzed (Participants) | 1 | 0
  02-003 - Total Staph/Week 4 | 6.70 |
  Subject 02-004 - Total Staphylococci/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-004 - Total Staphylococci/Pre |  | 5.15
  02-004 - Total Staph/Post: number analyzed (Participants) | 0 | 1
  02-004 - Total Staph/Post |  | 3.25
  02-004 - Total Staph/Week 4: number analyzed (Participants) | 0 | 1
  02-004 - Total Staph/Week 4 |  | 7.55
  Subject 02-005 - Total Staphylococci/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-005 - Total Staphylococci/Pre |  | 8.37
  02-005 - Total Staph/Post: number analyzed (Participants) | 0 | 1
  02-005 - Total Staph/Post |  | 6.67
  02-005 - Total Staph/Week 4: number analyzed (Participants) | 0 | 1
  02-005 - Total Staph/Week 4 |  | 6.69
  Subject 02-007 - Total Staphylococci/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-007 - Total Staphylococci/Pre | 0.00 |
  02-007 - Total Staph/Post: number analyzed (Participants) | 1 | 0
  02-007 - Total Staph/Post | 0.00 |
  02-007 - Total Staph/Week 4: number analyzed (Participants) | 1 | 0
  02-007 - Total Staph/Week 4 | 3.93 |
  Subject 02-008 - Total Staphylococci/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-008 - Total Staphylococci/Pre |  | 7.24
  02-008 - Total Staph/Post: number analyzed (Participants) | 0 | 1
  02-008 - Total Staph/Post |  | 5.93
  02-008 - Total Staph/Week 4: number analyzed (Participants) | 0 | 1
  02-008 - Total Staph/Week 4 |  | 3.43
  Subject 02-009 - Total Staphylococci/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-009 - Total Staphylococci/Pre | 6.97 |
  02-009 - Total Staph/Post: number analyzed (Participants) | 1 | 0
  02-009 - Total Staph/Post | 4.64 |
  02-009 - Total Staph/Week 4: number analyzed (Participants) | 1 | 0
  02-009 - Total Staph/Week 4 | 8.47 |
  Subject 02-010 - Total Staphylococci/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-010 - Total Staphylococci/Pre | 7.05 |
  02-010 - Total Staph/Post: number analyzed (Participants) | 1 | 0
  02-010 - Total Staph/Post | 6.87 |
  02-010 - Total Staph/Week 4: number analyzed (Participants) | 1 | 0
  02-010 - Total Staph/Week 4 | 8.15 |
  Subject 02-001 - Total S. aureus/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-001 - Total S. aureus/Pre | 0.00 |
  02-001 - Total S. aureus/Post: number analyzed (Participants) | 1 | 0
  02-001 - Total S. aureus/Post | 0.00 |
  02-001 - Total S. aureus/Week 4: number analyzed (Participants) | 1 | 0
  02-001 - Total S. aureus/Week 4 | 0.00 |
  Subject 02-002 - Total S. aureus/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-002 - Total S. aureus/Pre |  | 0.00
  02-002 - Total S. aureus/Post: number analyzed (Participants) | 0 | 1
  02-002 - Total S. aureus/Post |  | 0.00
  02-002 - Total S. aureus/Week 4: number analyzed (Participants) | 0 | 1
  02-002 - Total S. aureus/Week 4 |  | 0.00
  Subject 02-003 - Total S. aureus/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-003 - Total S. aureus/Pre | 0.00 |
  02-003 - Total S. aureus/Post: number analyzed (Participants) | 1 | 0
  02-003 - Total S. aureus/Post | 0.00 |
  02-003 - Total S. aureus/Week 4: number analyzed (Participants) | 1 | 0
  02-003 - Total S. aureus/Week 4 | 6.58 |
  Subject 02-004 - Total S. aureus/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-004 - Total S. aureus/Pre |  | 0.00
  02-004 - Total S. aureus/Post: number analyzed (Participants) | 0 | 1
  02-004 - Total S. aureus/Post |  | 0.00
  02-004 - Total S. aureus/Week 4: number analyzed (Participants) | 0 | 1
  02-004 - Total S. aureus/Week 4 |  | 0.00
  Subject 02-005 - Total S. aureus/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-005 - Total S. aureus/Pre |  | 0.00
  02-005 - Total S. aureus/Post: number analyzed (Participants) | 0 | 1
  02-005 - Total S. aureus/Post |  | 0.00
  02-005 - Total S. aureus/Week 4: number analyzed (Participants) | 0 | 1
  02-005 - Total S. aureus/Week 4 |  | 0.00
  Subject 02-007 - Total S. aureus/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-007 - Total S. aureus/Pre | 0.00 |
  02-007 - Total S. aureus/Post: number analyzed (Participants) | 1 | 0
  02-007 - Total S. aureus/Post | 0.00 |
  02-007 - Total S. aureus/Week 4: number analyzed (Participants) | 1 | 0
  02-007 - Total S. aureus/Week 4 | 0.00 |
  Subject 02-008 - Total S. aureus/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-008 - Total S. aureus/Pre |  | 6.89
  02-008 - Total S. aureus/Post: number analyzed (Participants) | 0 | 1
  02-008 - Total S. aureus/Post |  | 5.49
  02-008 - Total S. aureus/Week 4: number analyzed (Participants) | 0 | 1
  02-008 - Total S. aureus/Week 4 |  | 0.00
  Subject 02-009 - Total S. aureus/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-009 - Total S. aureus/Pre | 0.00 |
  02-009 - Total S. aureus/Post: number analyzed (Participants) | 1 | 0
  02-009 - Total S. aureus/Post | 0.00 |
  02-009 - Total S. aureus/Week 4: number analyzed (Participants) | 1 | 0
  02-009 - Total S. aureus/Week 4 | 0.00 |
  Subject 02-010 - Total S. aureus/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-010 - Total S. aureus/Pre | 0.00 |
  02-010 - Total S. aureus/Post: number analyzed (Participants) | 1 | 0
  02-010 - Total S. aureus/Post | 0.00 |
  02-010 - Total S. aureus/Week 4: number analyzed (Participants) | 1 | 0
  02-010 - Total S. aureus/Week 4 | 0.00 |
  Subject 02-001 - Total Coliforms/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-001 - Total Coliforms/Pre | 6.83 |
  02-001 - Total Coliforms/Post: number analyzed (Participants) | 1 | 0
  02-001 - Total Coliforms/Post | 3.53 |
  02-001 - Total Coliforms/Week 4: number analyzed (Participants) | 1 | 0
  02-001 - Total Coliforms/Week 4 | 0.00 |
  Subject 02-002 - Total Coliforms/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-002 - Total Coliforms/Pre |  | 6.84
  02-002 - Total Coliforms/Post: number analyzed (Participants) | 0 | 1
  02-002 - Total Coliforms/Post |  | 5.58
  02-002 - Total Coliforms/Week 4: number analyzed (Participants) | 0 | 1
  02-002 - Total Coliforms/Week 4 |  | 4.68
  Subject 02-003 - Total Coliforms/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-003 - Total Coliforms/Pre | 0.00 |
  02-003 - Total Coliforms/Post: number analyzed (Participants) | 1 | 0
  02-003 - Total Coliforms/Post | 0.00 |
  02-003 - Total Coliforms/Week 4: number analyzed (Participants) | 1 | 0
  02-003 - Total Coliforms/Week 4 | 0.00 |
  Subject 02-004 - Total Coliforms/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-004 - Total Coliforms/Pre |  | 0.00
  02-004 - Total Coliforms/Post: number analyzed (Participants) | 0 | 1
  02-004 - Total Coliforms/Post |  | 0.00
  02-004 - Total Coliforms/Week 4: number analyzed (Participants) | 0 | 1
  02-004 - Total Coliforms/Week 4 |  | 4.23
  Subject 02-005 - Total Coliforms/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-005 - Total Coliforms/Pre |  | 6.50
  02-005 - Total Coliforms/Post: number analyzed (Participants) | 0 | 1
  02-005 - Total Coliforms/Post |  | 5.56
  02-005 - Total Coliforms/Week 4: number analyzed (Participants) | 0 | 1
  02-005 - Total Coliforms/Week 4 |  | 6.26
  Subject 02-007 - Total Coliforms/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-007 - Total Coliforms/Pre | 7.33 |
  02-007 - Total Coliforms/Post: number analyzed (Participants) | 1 | 0
  02-007 - Total Coliforms/Post | 4.99 |
  02-007 - Total Coliforms/Week 4: number analyzed (Participants) | 1 | 0
  02-007 - Total Coliforms/Week 4 | 4.57 |
  Subject 02-008 - Total Coliforms/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-008 - Total Coliforms/Pre |  | 7.75
  02-008 - Total Coliforms/Post: number analyzed (Participants) | 0 | 1
  02-008 - Total Coliforms/Post |  | 7.37
  02-008 - Total Coliforms/Week 4: number analyzed (Participants) | 0 | 1
  02-008 - Total Coliforms/Week 4 |  | 0.00
  Subject 02-009 - Total Coliforms/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-009 - Total Coliforms/Pre | 0.00 |
  02-009 - Total Coliforms/Post: number analyzed (Participants) | 1 | 0
  02-009 - Total Coliforms/Post | 0.00 |
  02-009 - Total Coliforms/Week 4: number analyzed (Participants) | 1 | 0
  02-009 - Total Coliforms/Week 4 | 0.00 |
  Subject 02-010 - Total Coliforms/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-010 - Total Coliforms/Pre | 7.14 |
  02-010 - Total Coliforms/Post: number analyzed (Participants) | 1 | 0
  02-010 - Total Coliforms/Post | 6.89 |
  02-010 - Total Coliforms/Week 4: number analyzed (Participants) | 1 | 0
  02-010 - Total Coliforms/Week 4 | 8.24 |
  Subject 02-001 - Total Pseudomonads/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-001 - Total Pseudomonads/Pre | 0.00 |
  02-001 - Total Pseudomonads/Post: number analyzed (Participants) | 1 | 0
  02-001 - Total Pseudomonads/Post | 0.00 |
  02-001 - Total Pseudomonads/Week 4: number analyzed (Participants) | 1 | 0
  02-001 - Total Pseudomonads/Week 4 | 0.00 |
  Subject 02-002 - Total Pseudomonads/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-002 - Total Pseudomonads/Pre |  | 0.00
  02-002 - Total Pseudomonads/Post: number analyzed (Participants) | 0 | 1
  02-002 - Total Pseudomonads/Post |  | 0.00
  02-002 - Total Pseudomonads/Week 4: number analyzed (Participants) | 0 | 1
  02-002 - Total Pseudomonads/Week 4 |  | 0.00
  Subject 02-003 - Total Pseudomonads/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-003 - Total Pseudomonads/Pre | 0.00 |
  02-003 - Total Pseudomonads/Post: number analyzed (Participants) | 1 | 0
  02-003 - Total Pseudomonads/Post | 0.00 |
  02-003 - Total Pseudomonads/Week 4: number analyzed (Participants) | 1 | 0
  02-003 - Total Pseudomonads/Week 4 | 0.00 |
  Subject 02-004 - Total Pseudomonads/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-004 - Total Pseudomonads/Pre |  | 5.89
  02-004 - Total Pseudomonads/Post: number analyzed (Participants) | 0 | 1
  02-004 - Total Pseudomonads/Post |  | 4.87
  02-004 - Total Pseudomonads/Week 4: number analyzed (Participants) | 0 | 1
  02-004 - Total Pseudomonads/Week 4 |  | 4.43
  Subject 02-005 - Total Pseudomonads/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-005 - Total Pseudomonads/Pre |  | 0.00
  02-005 - Total Pseudomonads/Post: number analyzed (Participants) | 0 | 1
  02-005 - Total Pseudomonads/Post |  | 0.00
  02-005 - Total Pseudomonads/Week 4: number analyzed (Participants) | 0 | 1
  02-005 - Total Pseudomonads/Week 4 |  | 0.00
  Subject 02-007 - Total Pseudomonads/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-007 - Total Pseudomonads/Pre | 0.00 |
  02-007 - Total Pseudomonads/Post: number analyzed (Participants) | 1 | 0
  02-007 - Total Pseudomonads/Post | 0.00 |
  02-007 - Total Pseudomonads/Week 4: number analyzed (Participants) | 1 | 0
  02-007 - Total Pseudomonads/Week 4 | 0.00 |
  Subject 02-008 - Total Pseudomonads/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-008 - Total Pseudomonads/Pre |  | 0.00
  02-008 - Total Pseudomonads/Post: number analyzed (Participants) | 0 | 1
  02-008 - Total Pseudomonads/Post |  | 0.00
  02-008 - Total Pseudomonads/Week 4: number analyzed (Participants) | 0 | 1
  02-008 - Total Pseudomonads/Week 4 |  | 0.00
  Subject 02-009 - Total Pseudomonads/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-009 - Total Pseudomonads/Pre | 0.00 |
  02-009 - Total Pseudomonads/Post: number analyzed (Participants) | 1 | 0
  02-009 - Total Pseudomonads/Post | 0.00 |
  02-009 - Total Pseudomonads/Week 4: number analyzed (Participants) | 1 | 0
  02-009 - Total Pseudomonads/Week 4 | 0.00 |
  Subject 02-010 - Total Pseudomonads/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-010 - Total Pseudomonads/Pre | 0.00 |
  02-010 - Total Pseudomonads/Post: number analyzed (Participants) | 1 | 0
  02-010 - Total Pseudomonads/Post | 0.00 |
  02-010 - Total Pseudomonads/Week 4: number analyzed (Participants) | 1 | 0
  02-010 - Total Pseudomonads/Week 4 | 0.00 |
  Subject 02-001 - Total Strep/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-001 - Total Strep/Pre | 0.00 |
  02-001 - Total Strep/Post: number analyzed (Participants) | 1 | 0
  02-001 - Total Strep/Post | 0.00 |
  02-001 - Total Strep/Week 4: number analyzed (Participants) | 1 | 0
  02-001 - Total Strep/Week 4 | 0.00 |
  Subject 02-002 - Total Strep/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-002 - Total Strep/Pre |  | 0.00
  02-002 - Total Strep/Post: number analyzed (Participants) | 0 | 1
  02-002 - Total Strep/Post |  | 0.00
  02-002 - Total Strep/Week 4: number analyzed (Participants) | 0 | 1
  02-002 - Total Strep/Week 4 |  | 0.00
  Subject 02-003 - Total Strep/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-003 - Total Strep/Pre | 0.00 |
  02-003 - Total Strep/Post: number analyzed (Participants) | 1 | 0
  02-003 - Total Strep/Post | 0.00 |
  02-003 - Total Strep/Week 4: number analyzed (Participants) | 1 | 0
  02-003 - Total Strep/Week 4 | 0.00 |
  Subject 02-004 - Total Strep/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-004 - Total Strep/Pre |  | 0.00
  02-004 - Total Strep/Post: number analyzed (Participants) | 0 | 1
  02-004 - Total Strep/Post |  | 0.00
  02-004 - Total Strep/Week 4: number analyzed (Participants) | 0 | 1
  02-004 - Total Strep/Week 4 |  | 0.00
  Subject 02-005 - Total Strep/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-005 - Total Strep/Pre |  | 0.00
  02-005 - Total Strep/Post: number analyzed (Participants) | 0 | 1
  02-005 - Total Strep/Post |  | 0.00
  02-005 - Total Strep/Week 4: number analyzed (Participants) | 0 | 1
  02-005 - Total Strep/Week 4 |  | 0.00
  Subject 02-007 - Total Strep/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-007 - Total Strep/Pre | 0.00 |
  02-007 - Total Strep/Post: number analyzed (Participants) | 1 | 0
  02-007 - Total Strep/Post | 0.00 |
  02-007 - Total Strep/Week 4: number analyzed (Participants) | 1 | 0
  02-007 - Total Strep/Week 4 | 0.00 |
  Subject 02-008 - Total Strep/Pre: number analyzed (Participants) | 0 | 1
  Subject 02-008 - Total Strep/Pre |  | 0.00
  02-008 - Total Strep/Post: number analyzed (Participants) | 0 | 1
  02-008 - Total Strep/Post |  | 0.00
  02-008 - Total Strep/Week 4: number analyzed (Participants) | 0 | 1
  02-008 - Total Strep/Week 4 |  | 0.00
  Subject 02-009 - Total Strep/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-009 - Total Strep/Pre | 0.00 |
  02-009 - Total Strep/Post: number analyzed (Participants) | 1 | 0
  02-009 - Total Strep/Post | 0.00 |
  02-009 - Total Strep/Week 4: number analyzed (Participants) | 1 | 0
  02-009 - Total Strep/Week 4 | 0.00 |
  Subject 02-010 - Total Strep/Pre: number analyzed (Participants) | 1 | 0
  Subject 02-010 - Total Strep/Pre | 0.00 |
  02-010 - Total Strep/Post: number analyzed (Participants) | 1 | 0
  02-010 - Total Strep/Post | 0.00 |
  02-010 - Total Strep/Week 4: number analyzed (Participants) | 1 | 0
  02-010 - Total Strep/Week 4 | 0.00 |

2. Secondary Outcome: Photograph Area Measurements to Determine Reduction in Wound Size
Description: a) Reduction in wound size for up to 12 weeks post-debridement Photographs of the wound site were taken to determine the reduction in wound size and to assess healing progression of the study wound. Standardization of images was ensured by the Eykona® Wound Measurement System that uses small sterile 'targets' placed on the study wound to set the focus and position of the camera thus eliminating inconsistency between images acquisition time points. The photographs are stored on a USB (Universal Serial Bus) flash drive which will be archived with the study files.
Time Frame: Visit 2 through Visit 8 (12 weeks)
Population: All treated subjects
Measure: Number; unit: cm^2
Arm/Group | WoundWand™ Debridement Device | Standard of Care Sharp Debridement
Number analyzed (Participants) | 5 | 4
cm^2
  Subject 02-001 Visit 2/Pre Debridement: number analyzed (Participants) | 1 | 0
  Subject 02-001 Visit 2/Pre Debridement | NA — Area measurement not reported by study site to Sponsor. |
  02-001 Visit 2/Post Debridement: number analyzed (Participants) | 1 | 0
  02-001 Visit 2/Post Debridement | 80.24 |
  02-001 Visit 3/Week 1: number analyzed (Participants) | 1 | 0
  02-001 Visit 3/Week 1 | 57.24 |
  02-001 Visit 4/Week 2: number analyzed (Participants) | 1 | 0
  02-001 Visit 4/Week 2 | 58.36 |
  02-001 Visit 5/Week 3: number analyzed (Participants) | 1 | 0
  02-001 Visit 5/Week 3 | 50.15 |
  02-001 Visit 6/Week 4: number analyzed (Participants) | 1 | 0
  02-001 Visit 6/Week 4 | 52.12 |
  02-001 Visit 7/Week 6: number analyzed (Participants) | 1 | 0
  02-001 Visit 7/Week 6 | 35.61 |
  02-001 Visit 7/Week 6 measurement 2: number analyzed (Participants) | 1 | 0
  02-001 Visit 7/Week 6 measurement 2 | 29.70 |
  02-001 Visit 8/Week 12: number analyzed (Participants) | 1 | 0
  02-001 Visit 8/Week 12 | 17.84 |
  Subject 02-002 Visit 2/Pre Debridement: number analyzed (Participants) | 0 | 1
  Subject 02-002 Visit 2/Pre Debridement |  | 41.80
  02-002 Visit 2/Post Debridement: number analyzed (Participants) | 0 | 1
  02-002 Visit 2/Post Debridement |  | NA — Area measurement not reported by study site to Sponsor.
  02-002 Visit 3/Week 1: number analyzed (Participants) | 0 | 1
  02-002 Visit 3/Week 1 |  | 53.59
  02-002 Visit 4/Week 2: number analyzed (Participants) | 0 | 1
  02-002 Visit 4/Week 2 |  | 30.03
  02-002 Visit 5/Week 3: number analyzed (Participants) | 0 | 1
  02-002 Visit 5/Week 3 |  | 40.08
  02-002 Visit 6/Week 4: number analyzed (Participants) | 0 | 1
  02-002 Visit 6/Week 4 |  | 31.73
  02-002 Visit 7/Week 6: number analyzed (Participants) | 0 | 1
  02-002 Visit 7/Week 6 |  | 37.43
  02-002 Visit 7/Week 6 measurement 2: number analyzed (Participants) | 0 | 1
  02-002 Visit 7/Week 6 measurement 2 |  | 33.99
  02-002 Visit 8/Week 12: number analyzed (Participants) | 0 | 1
  02-002 Visit 8/Week 12 |  | 22.79
  Subject 02-003 Visit 2/Pre Debridement: number analyzed (Participants) | 1 | 0
  Subject 02-003 Visit 2/Pre Debridement | 6.80 |
  02-003 Visit 2/Post Debridement: number analyzed (Participants) | 1 | 0
  02-003 Visit 2/Post Debridement | 9.34 |
  02-003 Visit 3/Week 1: number analyzed (Participants) | 1 | 0
  02-003 Visit 3/Week 1 | 6.25 |
  02-003 Visit 4/Week 2: number analyzed (Participants) | 1 | 0
  02-003 Visit 4/Week 2 | 6.29 |
  02-003 Visit 4/Week 2 measurement 2: number analyzed (Participants) | 1 | 0
  02-003 Visit 4/Week 2 measurement 2 | 9.18 |
  02-003 Visit 5/Week 3: number analyzed (Participants) | 1 | 0
  02-003 Visit 5/Week 3 | 2.88 |
  02-003 Visit 6/Week 4: number analyzed (Participants) | 1 | 0
  02-003 Visit 6/Week 4 | 3.05 |
  02-003 Visit 7/Week 6: number analyzed (Participants) | 1 | 0
  02-003 Visit 7/Week 6 | 3.99 |
  02-003 Visit 8/Week 12: number analyzed (Participants) | 1 | 0
  02-003 Visit 8/Week 12 | 1.43 |
  Subject 02-004 Visit 2/Pre Debridement: number analyzed (Participants) | 0 | 1
  Subject 02-004 Visit 2/Pre Debridement |  | 2.37
  02-004 Visit 2/Post Debridement: number analyzed (Participants) | 0 | 1
  02-004 Visit 2/Post Debridement |  | 0.59
  02-004 Visit 3/Week 1: number analyzed (Participants) | 0 | 1
  02-004 Visit 3/Week 1 |  | 1.25
  02-004 Visit 3/Week 1 measurement 2: number analyzed (Participants) | 0 | 1
  02-004 Visit 3/Week 1 measurement 2 |  | 1.35
  02-004 Visit 4/Week 2: number analyzed (Participants) | 0 | 1
  02-004 Visit 4/Week 2 |  | 1.02
  02-004 Visit 5/Week 3: number analyzed (Participants) | 0 | 1
  02-004 Visit 5/Week 3 |  | 1.84
  02-004 Visit 6/Week 4: number analyzed (Participants) | 0 | 1
  02-004 Visit 6/Week 4 |  | 2.41
  02-004 Visit 7/Week 6: number analyzed (Participants) | 0 | 1
  02-004 Visit 7/Week 6 |  | 0.42
  02-004 Visit 8/Week 12: number analyzed (Participants) | 0 | 1
  02-004 Visit 8/Week 12 |  | 0.33
  Subject 02-005 Visit 2/Pre Debridement: number analyzed (Participants) | 0 | 1
  Subject 02-005 Visit 2/Pre Debridement |  | 16.20
  02-005 Visit 2/Post Debridement: number analyzed (Participants) | 0 | 1
  02-005 Visit 2/Post Debridement |  | 28.74
  02-005 Visit 3/Week 1: number analyzed (Participants) | 0 | 1
  02-005 Visit 3/Week 1 |  | 19.53
  02-005 Visit 3/Week 1 measurement 2: number analyzed (Participants) | 0 | 1
  02-005 Visit 3/Week 1 measurement 2 |  | 19.98
  02-005 Visit 4/Week 2: number analyzed (Participants) | 0 | 1
  02-005 Visit 4/Week 2 |  | 23.67
  02-005 Visit 5/Week 3: number analyzed (Participants) | 0 | 1
  02-005 Visit 5/Week 3 |  | 22.16
  02-005 Visit 6/Week 4: number analyzed (Participants) | 0 | 1
  02-005 Visit 6/Week 4 |  | 21.40
  02-005 Visit 7/Week 6: number analyzed (Participants) | 0 | 1
  02-005 Visit 7/Week 6 |  | 34.06
  02-005 Visit 8/Week 12: number analyzed (Participants) | 0 | 1
  02-005 Visit 8/Week 12 |  | 26.56
  Subject 02-007 Visit 2/Pre Debridement: number analyzed (Participants) | 1 | 0
  Subject 02-007 Visit 2/Pre Debridement | 23.56 |
  02-007 Visit 2/Pre Debridement: number analyzed (Participants) | 1 | 0
  02-007 Visit 2/Pre Debridement | 25.87 |
  02-007 Visit 2/Post Debridement: number analyzed (Participants) | 1 | 0
  02-007 Visit 2/Post Debridement | NA — Area measurement not reported by study site to Sponsor. |
  02-007 Visit 3/Week 1: number analyzed (Participants) | 1 | 0
  02-007 Visit 3/Week 1 | 26.91 |
  02-007 Visit 4/Week 2: number analyzed (Participants) | 1 | 0
  02-007 Visit 4/Week 2 | 23.02 |
  02-007 Visit 5/Week 3: number analyzed (Participants) | 1 | 0
  02-007 Visit 5/Week 3 | 24.89 |
  02-007 Visit 6/Week 4: number analyzed (Participants) | 1 | 0
  02-007 Visit 6/Week 4 | 28.04 |
  02-007 Visit 7/Week 6: number analyzed (Participants) | 1 | 0
  02-007 Visit 7/Week 6 | NA — Subject did not attend Visit 7. |
  02-007 Visit 8/Week 12: number analyzed (Participants) | 1 | 0
  02-007 Visit 8/Week 12 | NA — Subject did not attend Visit 8. |
  Subject 02-008 Visit 2/Pre Debridement: number analyzed (Participants) | 0 | 1
  Subject 02-008 Visit 2/Pre Debridement |  | 29.53
  02-008 Visit 2/Post Debridement: number analyzed (Participants) | 0 | 1
  02-008 Visit 2/Post Debridement |  | 86.16
  02-008 Visit 3/Week 1: number analyzed (Participants) | 0 | 1
  02-008 Visit 3/Week 1 |  | 50.26
  02-008 Visit 3/Week 1 measurement 2: number analyzed (Participants) | 0 | 1
  02-008 Visit 3/Week 1 measurement 2 |  | 85.47
  02-008 Visit 4/Week 2: number analyzed (Participants) | 0 | 1
  02-008 Visit 4/Week 2 |  | 30.13
  02-008 Visit 4/Week 2 measurement 2: number analyzed (Participants) | 0 | 1
  02-008 Visit 4/Week 2 measurement 2 |  | 72.20
  02-008 Visit 5/Week 3: number analyzed (Participants) | 0 | 1
  02-008 Visit 5/Week 3 |  | 19.65
  02-008 Visit 5/Week 3 measurement 2: number analyzed (Participants) | 0 | 1
  02-008 Visit 5/Week 3 measurement 2 |  | 33.32
  02-008 Visit 6/Week 4: number analyzed (Participants) | 0 | 1
  02-008 Visit 6/Week 4 |  | 93.46
  02-008 Visit 6/Week 4 measurement 2: number analyzed (Participants) | 0 | 1
  02-008 Visit 6/Week 4 measurement 2 |  | 24.75
  02-008 Visit 7/Week 6: number analyzed (Participants) | 0 | 1
  02-008 Visit 7/Week 6 |  | NA — Subject did not attend Visit 7.
  02-008 Visit 8/Week 12: number analyzed (Participants) | 0 | 1
  02-008 Visit 8/Week 12 |  | NA — Subject did not attend Visit 8.
  Subject 02-009 Visit 2/Pre Debridement: number analyzed (Participants) | 1 | 0
  Subject 02-009 Visit 2/Pre Debridement | 50.49 |
  02-009 Visit 2/Post Debridement: number analyzed (Participants) | 1 | 0
  02-009 Visit 2/Post Debridement | 35.05 |
  02-009 Visit 3/Week 1: number analyzed (Participants) | 1 | 0
  02-009 Visit 3/Week 1 | 67.80 |
  02-009 Visit 4/Week 2: number analyzed (Participants) | 1 | 0
  02-009 Visit 4/Week 2 | 26.84 |
  02-009 Visit 5/Week 3: number analyzed (Participants) | 1 | 0
  02-009 Visit 5/Week 3 | 23.02 |
  02-009 Visit 6/Week 4: number analyzed (Participants) | 1 | 0
  02-009 Visit 6/Week 4 | 38.27 |
  02-009 Visit 7/Week 6: number analyzed (Participants) | 1 | 0
  02-009 Visit 7/Week 6 | NA — Subject did not attend Visit 7. |
  02-009 Visit 8/Week 12: number analyzed (Participants) | 1 | 0
  02-009 Visit 8/Week 12 | NA — Subject did not attend Visit 8. |
  Subject 02-010 Visit 2/Pre Debridement: number analyzed (Participants) | 1 | 0
  Subject 02-010 Visit 2/Pre Debridement | 9.03 |
  02-010 Visit 2/Post Debridement: number analyzed (Participants) | 1 | 0
  02-010 Visit 2/Post Debridement | 9.39 |
  02-010 Visit 3/Week 1: number analyzed (Participants) | 1 | 0
  02-010 Visit 3/Week 1 | 24.15 |
  02-010 Visit 3/Week 1 measurement 2: number analyzed (Participants) | 1 | 0
  02-010 Visit 3/Week 1 measurement 2 | 6.55 |
  02-010 Visit 4/Week 2: number analyzed (Participants) | 1 | 0
  02-010 Visit 4/Week 2 | 6.99 |
  02-010 Visit 5/Week 3: number analyzed (Participants) | 1 | 0
  02-010 Visit 5/Week 3 | 5.08 |
  02-010 Visit 6/Week 4: number analyzed (Participants) | 1 | 0
  02-010 Visit 6/Week 4 | 15.42 |
  02-010 Visit 7/Week 6: number analyzed (Participants) | 1 | 0
  02-010 Visit 7/Week 6 | NA — Area measurement not reported by study site to Sponsor. |
  02-010 Visit 8/Week 12: number analyzed (Participants) | 1 | 0
  02-010 Visit 8/Week 12 | NA — Area measurement not reported by study site to Sponsor. |

3. Secondary Outcome: Wound Status Using Bates-Jensen Wound Assessment - Total Score
Description: The Bates-Jensen Wound Assessment Tool is a 13-item questionnaire (size, depth, edges, undermining, necrotic tissue type, exudate type, exudate amount, skin color surrounding wound, peripheral tissue edema, peripheral tissue induration, granulation tissue, epithelialization) used to assess wound status.
  Total score is determined by adding together the sub-scores from each of the 13 items, with a higher score indicating a more severe wound status. Each of the 13 item scores ranged from 1 to 5 possible points. Minimum score of 13 indicated the best outcome, maximum score of 65 indicated the worst outcome.
Time Frame: Screening through Visit 8 (12 weeks)
Population: All subjects seen and assessed at each time point.
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | WoundWand™ Debridement Device | Standard of Care Sharp Debridement
Number analyzed (Participants) | 5 | 4
total score on a scale
  Visit 1/Screening | 33.2 (3.1) | 33.8 (4.8)
  Visit 2/Debridement | 35.2 (5.8) | 33.3 (5.6)
  Visit 3/Week 1 | 31.0 (6.4) | 34.0 (5.0)
  Visit 4/Week 2 | 27.8 (2.9) | 33.3 (5.4)
  Visit 5/Week 3 | 25.2 (3.1) | 33.3 (6.1)
  Visit 6/Week 4: number analyzed (Participants) | 4 | 4
  Visit 6/Week 4 | 25.5 (5.7) | 32.3 (7.6)
  Visit 7/Week 6: number analyzed (Participants) | 3 | 3
  Visit 7/Week 6 | 18.7 (0.6) | 31.0 (10.1)
  Visit 8/Week 12: number analyzed (Participants) | 3 | 3
  Visit 8/Week 12 | 16.0 (1.7) | 31.0 (20.9)

4. Secondary Outcome: Braden Scale for Predicting Pressure Sore Risk - Total Score
Description: The Braden Scale, performed by the Investigator (or designee), is a 6-item questionnaire (sensory perception, moisture, activity, mobility, nutrition, and friction &shear) used to assess the subject's level of risk for development of pressure ulcers.
  Total score is determined by adding together the sub-scores from each of the 6 items, with a lower score indicating a higher risk for developing pressure ulcers.
  Braden Scale thresholds:
  19-23 = not at risk 15-18 = preventative interventions 13-14 = moderate risk 10-12 = high risk 6-9 = very high risk
  Sub-score ranges:
  Sensory perception: 1 - 4 Moisture: 1 - 4 Activity: 1 - 4 Mobility: 1 - 4 Nutrition: 1 - 4 Friction & Shear: 1 - 3
  Total score minimum of 6 indicated a very high risk outcome, maximum score of 23 indicated the subject not at risk.
Time Frame: Screening through Visit 8 (12 weeks)
Population: All available subjects at each time point.
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | WoundWand™ Debridement Device | Standard of Care Sharp Debridement
Number analyzed (Participants) | 5 | 4
total score on a scale
  Visit 1/Screening | 17.8 (2.6) | 18.5 (3.1)
  Visit 3/Week 1 | 17.6 (2.9) | 18.0 (2.2)
  Visit 4/Week 2 | 17.8 (3.1) | 18.0 (2.2)
  Visit 5/Week 3 | 17.8 (3.6) | 18.3 (2.9)
  Visit 6/Week 4 | 17.8 (2.8) | 18.5 (3.3)
  Visit 7/Week 6: number analyzed (Participants) | 3 | 3
  Visit 7/Week 6 | 18.0 (1.7) | 20.0 (4.4)
  Visit 8/Week 12: number analyzed (Participants) | 3 | 3
  Visit 8/Week 12 | 19.3 (3.8) | 20.0 (4.4)

ADVERSE EVENTS:
Time Frame: AEs were collected from the time of enrollment until study completion at 12 weeks post debridement, study withdrawal, or study termination, whichever came first.
Groups:
- WoundWand™ Debridement Device: Group I - Coblator IQTM Controller plus WoundWand™ Debridement Device. Electrical energy that removes necrotic, ischemic, and/or infected tissue within a wound.
  WoundWand™ Debridement Device: Group I - Electrical energy that removes necrotic, ischemic, and/or infected tissue within a wound
Arm/Group | WoundWand™ Debridement Device | Standard of Care Sharp Debridement
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 4/5 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WoundWand™ Debridement Device (N=5) | Standard of Care Sharp Debridement (N=4)
2:1 AV block and bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Micro groin wound infection (Infections and infestations) | 1 (1) | 0 (0)
Infection to wound (Infections and infestations) | 0 (0) | 1 (1)
Chronic wound (Infections and infestations) | 2 (2) | 1 (1)
Infection to foot ulcer (Infections and infestations) | 1 (1) | 0 (0)
Serratia growth on bone (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated due to lower than anticipated accrual rate and the desire to reassess overall study strategy; therefore, statistically sound conclusions regarding safety, effectiveness, and risk/benefit profile of the device can't be made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes